CLINICAL TRIAL: NCT06693856
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study on the Efficacy and Safety of Different Methylprednisolone Pulse Therapy Regimens for the Treatment of Graves' Ophthalmopathy
Brief Title: Multi-center Prospective Clinical Study on Glucocorticoid Pulse Therapy for Graves' Ophthalmopathy (GO)
Acronym: GO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zou Junjie (Other)
Responsible Party: Sponsor-Investigator, Zou Junjie, Professor, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024SL126
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves ophthalmopathy, methylprednisolone, therapy regimens
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- a high-dose group (Active Comparator): methylprednisolone 500mg, D1-3, once every 4 weeks
  Interventions: Drug: High-Dose Methylprednisolone
- a low-dose group (Experimental): methylprednisolone 1mg/kg, D1-3, once every 4 weeks
  Interventions: Drug: Low-Dose Methylprednisolone

INTERVENTIONS:
Drug: High-Dose Methylprednisolone — Methylprednisolone 500mg, administered intravenously once daily for 3 consecutive days, repeated every 4 weeks for a total of 24 weeks, followed by a follow-up period.
  Arms: a high-dose group
Drug: Low-Dose Methylprednisolone — Methylprednisolone is administered at a dose of 1mg/kg, given as an intravenous injection once daily for 3 consecutive days, repeated every 4 weeks for a total of 24 weeks, followed by a follow-up period.
  Arms: a low-dose group

SUMMARY:
This study plans to include newly diagnosed, active, moderate to severe Graves' ophthalmopathy patients, divided into a high-dose group (methylprednisolone 500mg, D1-3, once every 4 weeks) and a low-dose group (methylprednisolone 1mg/kg, D1-3, once every 4 weeks), with a treatment duration of 24 weeks to compare the efficacy and safety of the two groups. Additionally, this study will extend the follow-up to 48 weeks to observe the recurrence rate after treatment in both groups, exploring the heterogeneity of the active course of Graves' ophthalmopathy.

DETAILED DESCRIPTION:
Graves' ophthalmopathy (GO) is an organ-specific autoimmune disease closely related to the thyroid gland, typically manifested by proptosis, eyelid swelling, eye pain, and double vision. Mild GO may resolve with the control of hyperthyroidism, while moderate to severe GO can severely damage vision and require more aggressive treatment. Glucocorticoids are the first-line treatment for moderate to severe, active GO, and intravenous methylprednisolone is more effective than oral glucocorticoids. The 2021 clinical practice guidelines of the European Group on Graves' Orbitopathy (EUGOGO) recommend that the optimal dosage regimen for methylprednisolone is once a week for 12 weeks, with a cumulative dose of 4.5 grams. For the most severe cases, a higher cumulative dose of up to 8 grams can also be used as monotherapy.

Starting from the 1990s, the Endocrinology Department of Shanghai Changzheng Hospital began to admit patients with Graves' ophthalmopathy and initiated immunosuppressive pulse therapy, accumulating nearly 1000 cases of GO, making it the hospital with the most patients with Graves' ophthalmopathy in Shanghai and even nationwide. The monthly pulse therapy regimen has a high treatment response rate, a low relapse rate, and good safety. However, there are still a series of unresolved issues with glucocorticoid pulse therapy for Graves' ophthalmopathy. Firstly, the optimal cumulative dose of methylprednisolone has not been established. Secondly, the active course of Graves' ophthalmopathy varies greatly among individuals, with reports ranging from a few months to several years, and the pulse therapy has not yet been individualized. Thirdly, there is a significant difference in individual sensitivity to glucocorticoids; the fixed high-dose administration of methylprednisolone at 500mg per session lacks sufficient evidence. Calculating the single-dose administration based on body weight or surface area may be more reasonable.

The efficacy and safety of different dosage regimens of methylprednisolone pulse therapy for Graves' ophthalmopathy will be further explored. This study plans to include newly diagnosed, active, moderate to severe Graves' ophthalmopathy patients, divided into a high-dose group (methylprednisolone 500mg, D1-3, once every 4 weeks) and a low-dose group (methylprednisolone 1mg/kg, D1-3, once every 4 weeks), with a treatment duration of 24 weeks to compare the efficacy and safety of the two groups. Additionally, this study will extend the follow-up to 48 weeks to observe the recurrence rate after treatment in both groups, exploring the heterogeneity of the active course of Graves' ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily accept the study and sign the informed consent form.
2. Age between 25 and 70 years old at the time of enrollment, both males and females are eligible.
3. Newly diagnosed Graves' ophthalmopathy, moderate to severe active patients. The criteria for moderate to severe GO are: ① eyelid retraction ≥2mm; ② moderate to severe involvement of orbital soft tissues; ③ proptosis ≥20mm; ④ periodic or persistent diplopia. Meeting one of the above four criteria is sufficient.

   The criteria for active GO are: CAS score ≥4 points. Scoring criteria: ① spontaneous retro-ocular pain; ② pain on eye movement; ③ conjunctival congestion; ④ eyelid congestion; ⑤ chemosis of the conjunctiva; ⑥ swelling of the caruncle; ⑦ eyelid edema. One point is recorded for each of the above seven symptoms if present, and zero if absent.
4. The onset of Graves' ophthalmopathy does not exceed 12 months, and those who have not been treated with glucocorticoids or other immunosuppressive agents.
5. Women of childbearing age must use effective contraceptive measures.
6. At the time of screening, hyperthyroidism in the study subjects should be basically controlled. Thyroid function should be normal or only mildly abnormal, defined as FT4 and FT3 levels within 50% of the upper and lower limits of the normal range. Mild thyroid dysfunction should be corrected as much as possible, and a normal thyroid function state should be maintained throughout the clinical trial period.

Exclusion Criteria:

1. Pregnant women, women who are breastfeeding, or women planning to become pregnant during the trial period.
2. Severe cardiac diseases such as myocardial infarction, unstable angina, and chronic heart failure.
3. Known liver diseases, or alanine transaminase (ALT) levels more than 1.5 times the upper limit of normal.
4. Chronic kidney disease, or serum creatinine >135 umol/L (>1.5 mg/dL).
5. Individuals with diabetes, and HbA1c >9.0%.
6. Individuals with a history of alcohol abuse or drug use.
7. Subjects with a white blood cell count <4.0×10^9/L, or a platelet count <80×10^9/L.
8. Significant anemia (hemoglobin levels <110 g/L in males, <100 g/L in females).
9. Patients with psychiatric disorders, or those who are non-cooperative.
10. Individuals with optic nerve involvement requiring orbital decompression surgery. Defined as a decrease in vision by more than two lines in the past six months, or new visual field defects, or color vision deficiencies.
11. Corneal ulcers, contraindications for glucocorticoid treatment.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate, ORR | From enrollment to the end of treatment at 24 weeks
  The percentage of subjects with improvement in Graves' ophthalmopathy at week 24.

SECONDARY OUTCOMES:
CAS and proptosis | From enrollment to the end of treatment at 24 weeks
  To assess the percentage of subjects in the high-dose group and the low-dose group at week 24 who have a reduction of ≥2 points in CAS (Clinical Activity Score) and a reduction of ≥2mm in proptosis compared to baseline, provided that there is no corresponding worsening in the contralateral eye (increase in CAS of ≥2 points or increase in proptosis of ≥2mm).
Clinical Activity Score | From enrollment to the end of treatment at 24 weeks
  To assess the percentage of subjects in the high-dose group and the low-dose group at week 24 who have a CAS of 0 or 1 in the study eye.
proptosis | From enrollment to the end of treatment at 24 weeks
  To assess the mean change in proptosis of the study eye from baseline to week 24 in the high-dose group and the low-dose group.

OTHER OUTCOMES:
Recurrence Rate, RR | From enrollment to the end of treatment at 48 weeks
  The percentage of subjects with Graves' ophthalmopathy worsening again at week 48 compared to week 24 in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zou JJ Professor, Principal Investigator — Shanghai Changzheng Hospital
Locations (3):
- China (3):
  - Shanghai Changzhen Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Longhua Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The shared data will include, but not be limited to, the participants' baseline characteristics, clinical measurements, medical history, clinical laboratory results, adverse events, as well as randomization results and treatment outcomes. Data will only be provided after application and approval.
Supporting Information: Analytic Code
Time Frame: The IPD and supporting information will be available starting from July 1, 2027 for 6 months.
Access Criteria: Data will only be provided after application and approval. Applicants must provide a reasonable data usage plan and commit to protecting participant privacy. Data usage must comply with relevant ethical and legal requirements. Interested researchers need to submit data sharing requests through the designated Clinical Trial Management Public Platform. Requests will be reviewed by the platform's management committee. Once approved, researchers will be granted access to de-identified IPD. The data will be stored on the servers of the Clinical Trial Management Public Platform, and the access address is: http://www.medresman.org.cn/login.aspx.